CLINICAL TRIAL: NCT01448694
Title: Non-invasive Hemodynamic Monitoring During Blood Donation for Developing Models of Early Blood Loss.
Status: Completed | Type: Observational
Sponsor: University of Colorado, Denver (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: 10-1421
Record Dates: First submitted 2011-10-05; First posted 2011-10-07 (Estimated); Last update posted 2014-12-03 (Estimated); Status verified 2014-12

CONDITIONS: Hemorrhage
Keywords: Hemorrhage
MeSH Terms: conditions — Hemorrhage

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Blood donors: Healthy volunteers who are donating a pint of whole blood
  Interventions: Other: No treatment

INTERVENTIONS:
Other: No treatment — No treatment, only collecting observational data.

SUMMARY:
This study is part of a Phase II STTR project to develop an algorithm called CipherSensor to apply feature extraction and machine learning techniques to non-invasive hemodynamic data to identify early signs of acute blood loss. The availability of this information may help to establish required interventions for treating trauma patients and battlefield casualties.

Study hypothesis: Hemodynamic changes measured non-invasively during the blood donation process can be modeled to provide early estimations of blood loss.

ELIGIBILITY:
Inclusion Criteria:

* Approved by Children's Hospital Colorado Blood Donation Center for blood donation
* Age 18 -89 years
* Previously donated blood (lower likelihood of vasovagal response)

Exclusion Criteria:

* Pregnant
* Incarcerated
* Limited access to or compromised monitoring sites for non-invasive sensors: finger, ear and forehead sensors, oral/nasal cannula, 3 ECG electrodes.

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy adults
Sampling Method: Non-Probability Sample
Enrollment: 320 (Actual)
Dates: Start 2011-11; Primary Completion 2013-10 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Algorithm | 24 months
  Mathematical model of early blood loss

CONTACTS AND LOCATIONS:
Overall Officials: Steve Moulton, MD, Principal Investigator — Children's Hospital Colorado
Locations (1):
- Children's Hospital Colorado, Aurora, Colorado, United States